CLINICAL TRIAL: NCT07203781
Title: Unraveling PEEP-induced Effects on Respiratory dRivE and EFfort in Acute Hypoxemic Respiratory Failure: the REEF Study
Brief Title: PEEP-induced Effects on Respiratory dRivE and EFfort
Acronym: REEF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Università Cattolica del Sacro Cuore, Rome, Italy (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NL-009995
Record Dates: First submitted 2025-09-04; First posted 2025-10-02 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-09

CONDITIONS: ARDS (Moderate or Severe); Acute Hypoxemic Respiratory Failure
Keywords: PEEP; effort; drive; PSV; pressure support ventilation; AHRF; ARDS; diaphragm; NME
MeSH Terms: conditions — Lymphoma, Follicular; Respiratory Insufficiency

STUDY DESIGN:
Intervention Model Description: Interventional, prospective physiological study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental)
  Interventions: Other: PEEP level changes

INTERVENTIONS:
Other: PEEP level changes — For each patient, six different PEEP levels (15-12-10-8-5-2 cmH2O) will be tested during a decremental PEEP trial. During each step, neural respiratory drive, inspiratory effort, expiratory muscle activity, lung inflation pattern through electrical impedance tomography, respiratory muscle geometry and function through ultrasound and surface EMG, gas exchange and hemodynamics data will be collected.

SUMMARY:
Rationale:

In patients with acute hypoxemic respiratory failure (AHRF), preserving spontaneous breathing during mechanical ventilation offers physiological benefits, but also carries risks. While spontaneous breathing improves gas exchange and limits diaphragm atrophy, strong inspiratory efforts may worsen lung and diaphragm injury. Balancing these factors requires refined and tailored strategies, such as the modulation of PEEP. However, the impact of PEEP on neural respiratory drive and inspiratory effort is very heterogenous, and these two entities have only been studied separately in limited subsets of patients and healthy subjects. Additionally, it remains unclear whether the major determinant of PEEP-induced changes in respiratory drive and effort is represented by variations in diaphragm geometry, lung compliance, or by the presence of expiratory muscles recruitment, which may counteract its effect.

Objective:

The primary objective is to determine the effect of PEEP on diaphragm neuromechanical efficiency (i.e. an index of neural respiratory drive and inspiratory effort) in patients with acute hypoxemic respiratory failure during invasive assisted mechanical ventilation. The secondary objective is to determine the major physiological contributors to PEEP-mediated changes in diaphragm neuromechanical efficiency.

Study design: Prospective, physiological study. Study population: Invasively mechanically ventilated adult patients admitted to the ICU.

Intervention:

For each patient, six different PEEP levels (15-12-10-8-5-2 cmH2O) will be tested during a decremental PEEP trial. During each step, neural respiratory drive, inspiratory effort, expiratory muscle activity, lung inflation pattern through electrical impedance tomography, respiratory muscle geometry and function through ultrasound and surface EMG, gas exchange and hemodynamics data will be collected.

Main study parameters/endpoints:

The primary outcome of the study will be the evaluation of PEEP-mediated changes in diaphragm neuromechanical efficiency (NME).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Acute hypoxemic respiratory failure (AHRF) with a PaO2/FiO2-ratio ≤ 200
* Patient on invasive assisted mechanical ventilation in pressure support mode exhibiting valid inspiratory efforts (occlusion pressure > 5 cmH2O).

Exclusion Criteria:

* Pre-existent neuromuscular disease
* History of chronic respiratory failure requiring long-term oxygen therapy
* Muscle paralysis
* Pneumothorax
* Contra-indication to EIT monitoring (e.g. burns, pacemaker, thoracic wounds limiting electrode placement)
* Contra-indications for EAdi or oesophageal balloon catheter placement (e.g. history of gastric bypass surgery, gastro-oesophageal junction surgery, oesophageal stricture, recent upper gastrointestinal hemorrhage or known/suspected varices).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-09-02 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
PEEP-related changes in diaphragm neuromechanical efficiency (NME) | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  The primary endpoint of this study will be the evaluation of PEEP-induced changes in diaphragm neuromechanical efficiency (NME, cmH2O/µV), calculated as the ratio between the change in transdiaphragmatic pressure (representing inspiratory effort in cmH2O and assessed through the use of esophageal and gastric manometry) and the change in diaphragm electrical activity (neural respiratory drive, expressed in µV and measured through diaphragm EMG by a dedicated nasogastric tube) for each inspiration (ΔPdi/ΔEAdi). NME is an index of diaphragm efficiency and of potential electromechanical uncoupling, a key PEEP-mediated effect on the diaphragm. Its assessment combines changes in neural respiratory drive and inspiratory effort after a change in PEEP, which will be assessed individually and combined as a ratio as primary outcome.

SECONDARY OUTCOMES:
PEEP-induced changes in inspiratory effort | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Inspiratory effort will be assessed through esophageal pressure monitoring and expressed in cmH2O.
PEEP-induced changes in neural respiratory drive | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Neural respiratory drive will be assessed through the monitoring of the electrical activity of the diaphragm, performed with the use of a dedicated nasogastric tube equipped with electrodes and expressed in µV.
PEEP-induced effects on partitioned respiratory system mechanics | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Respiratory mechanics assessed through ventilator and esophageal/gastric manometry, inlcuding end-expiratory, end-inspiratory and driving transpulmonary pressure (expressed in cmH2O).
PEEP induced effects on tidal volume | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Changes in expired tidal volume will be monitored from the ventilator (expressed in mL)
PEEP-induced effects on end-expiratory lung impedance | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  End-expiratory lung impedance will be assessed with electrical impedance tomography (EIT) and expressed in arbitrary units and as percentage change from baseline.
PEEP-induced effects on amount of pendelluft | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Pendelluft will be examined through electrical impedance tomography monitoring and expressed as % of total tidal impedance variation.
PEEP-induced changes in diaphragm thickening fraction assessed through ultrasound | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected once within the last 10 minutes of each step.
  Diaphragm thickening fraction will be assessed and expressed in %, through the formula: (End-inspiratory thickness - End-expiratory thickness) / End-expiratory thickness × 100.
PEEP-induced effects on internal oblique muscle thickening fraction | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected once within the last 10 minutes of each step.
  Internal oblique muscle thickening fraction will be measured through ultrasound and expressed in %, with the following formula: (End-inspiratory thickness - End-expiratory thickness) / End-expiratory thickness × 100.
PEEP-induced changes in gastric pressure during expiration | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Expiratory muscle activity will be assessed through monitoring of gastric pressure swings during expiration and expressed in cmH2O.
PEEP-induced changes in abdominal wall muscles expiratory activity | Measurements will be conducted throughout the protocol at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected recording the last 10 minutes of each step.
  Abdominal wall muscles expiratory activity will be assessed and quantified through the use of surface EMG of the abdominal wall, and expressed in µV.
PEEP-induced effects on gas exchange | Measurements will be conducted throughout the protocol at baseline and at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected once in the last 10 minutes of each step.
  Effects on gas exchange, including PaO2 and PaCO2 monitoring (mmHg), will be evaluated through arterial blood gas monitoring.
PEEP-induced effects on arterial blood pressure | Measurements will be conducted throughout the protocol at baseline and at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected once in the last 10 minutes of each step.
  Hemodynamics will be assessed through standard invasive blood pressure and will include the recording of systolic, diastolic and mean arterial blood pressure (mmHg).
PEEP-induced effects on heart rate | Measurements will be conducted throughout the protocol at baseline and at each of the 6 PEEP levels tested: 15, 12, 10, 8, 5 and 2 cmH2O. Each PEEP step will last 30 minutes, and measurements will be collected once in the last 10 minutes of each step.
  Heart rate will be monitored and expressed in beats per minute.

CONTACTS AND LOCATIONS:
Overall Officials: Jonne Doorduin, PhD, Principal Investigator — Radboud University Medical Center; Leo Heunks, M.D., PhD, Study Chair — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided